CLINICAL TRIAL: NCT05762809
Title: Kinesiophobia After Anterior Cruciate Ligament Reconstruction.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TUHST-1
Record Dates: First submitted 2023-02-16; First posted 2023-03-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Kinesiophobia; ACL Injury
MeSH Terms: conditions — Kinesiophobia; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kinesiophobia tests (Experimental): Patients were assessed using the Tampa Scale of Kinesiophobia (TSK-17), Knee injury and Osteoarthritis Outcome Score (KOOS), and Oxford Knee score (OKS). Ten minutes cycling with light resistance on a stationary bike was used for warm up before the physical tests. Quadriceps and hamstring muscle isokinetic strength was assessed at 60°/sec and 180°/sec using a Humac Norm Isokinetic dynamometer (Stoughton, United States). Functional performance was tested with the single-leg hop test for distance and the Y-balance test for anterior reach. The non-operated leg was tested first. All physical tests were supervised by the same specialized physiotherapists.
  Interventions: Diagnostic Test: Tampa Scale of Kinesiophobia (TSK-17); Diagnostic Test: Knee injury and Osteoarthritis Outcome Score (KOOS); Diagnostic Test: Oxford Knee Score (OKS) scoring; Diagnostic Test: Quadriceps and hamstring muscle isokinetic strength; Diagnostic Test: Single-leg hop test; Diagnostic Test: Y-balance test; Diagnostic Test: Anthropometric measurements

INTERVENTIONS:
Diagnostic Test: Tampa Scale of Kinesiophobia (TSK-17) — The Tampa Scale of Kinesiophobia (TSK-17) was developed as a self-reported checklist to measure fear of pain during movement and fear of reinjury. The TSK-17 consists of 17 questions. Standardized answer options are given as a 4-point Likert scale, and each question is assigned a score from 1 to 4. A normalized score between 17 and 68 points is calculated. A score of 37 or over indicates kinesiophobia.
Diagnostic Test: Knee injury and Osteoarthritis Outcome Score (KOOS) — The KOOS consists of five subscales - Symptoms (S), Pain (P), Functional activities of daily living (ADL), Sport and Recreation Function (Sport/Rec) and Knee-Related Quality of life (QOL) - and total KOOS Outcome (O) scores. Standardized answer options are provided (5 Likert boxes), and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Diagnostic Test: Oxford Knee Score (OKS) scoring — OKS consists of 12 questions. Standardized answer options are provided (5 Likert boxes), and each question is assigned a score from 0 to 4. A score of 40-48 indicates no symptoms or satisfactory joint function, 30-39 moderate knee arthritis, 20-29 moderate to severe knee arthritis, and 0-19 severe knee arthritis.
Diagnostic Test: Quadriceps and hamstring muscle isokinetic strength — Quadriceps and hamstring muscle strength at 60˚/s and 180˚/s were measured with an isokinetic dynamometer. For 180˚/s, five trial and fifteen testing repetitions were used, and for 60˚/s, three trial and three testing repetitions were used. The resting time between trial and testing was two minutes, between different speeds one minute, and between legs two minutes. The maximum peak torques were used in the statistical analysis.
Diagnostic Test: Single-leg hop test — The single-leg hop test (SLHT) for distance was used for lower limb functional testing. The test started with the participant standing on one leg, toes behind a marked line, and hands on hips throughout to avoid aiding the jump by swinging the arms. The participant was instructed to jump as far as possible and land on the same leg without losing balance. If the patient made contact with the ground with the contralateral limb, lost balance, or made additional hops after landing, the distance was not measured and the jump void. The distance was measured from the starting line to the heel of the leg being tested. For both legs, three trials and three jumps for maximal effort were allowed. The longest distance for both the left leg and the right leg were used in the statistical analysis.
Diagnostic Test: Y-balance test — The Y-balance test (YBT) (Move2Perform, United States) for anterior reach was used to measure dynamic balance. Participants performed three trials to familiarize themselves with the test, and then undertook three tests. The test started with the participant standing barefoot on the testing kit. The patients had to push a wooden box with the contralateral leg as far as possible with continuous movement and return to their starting position without losing balance. The longest distance achieved was used in the statistical analysis.
Diagnostic Test: Anthropometric measurements — Body mass (kg) and height (cm) were measured, and the body mass index (BMI) was calculated as kg/m2.

SUMMARY:
Anterior cruciate ligament (ACL) rupture is a serious trauma with long-term consequences to the athlete. Psychological and physiological factors may negatively affect patient recovery and increase reinjury rate after anterior cruciate ligament reconstruction (ACLR), and development of kinesiophobia is also possible.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) rupture is a serious trauma with long-term consequences to the athlete. Return to sports at the pre-injury level after anterior cruciate ligament reconstruction (ACLR) is reported between 55 and 83%. Psychological and physiological factors can negatively affect patient recovery and increase reinjury rate after ACLR. In daily practice, surgeons and physiotherapists see athletes struggling to improve muscle strength and complaining of a lack of self-confidence and fear of reinjury during their progress to return to sports.

Kinesiophobia in ACLR patients is used to determine fear of pain, lack of self-confidence, and fear of reinjury. Patients with self-reported fear are less active, have decreased muscle function, and increased risk of a second ACL injury. Lower rates of return to sports are reported in athletes with kinesiophobia after ACLR. To measure kinesiophobia, the self-reported Tampa Scale of Kinesiophobia (TSK-17) test is widely used. The original TSK was developed and described by Miller et al. in 1991. In ACLR patients, the risk of developing fear was previously measured in a large systematic review of 2175 patients, in which 514 (24%) reported a psychological reason for not returning to sports.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent ACLR by three orthopaedic surgeons at the Tartu University Hospital Sports Traumatology Centre between 2013 and 2019.

Exclusion Criteria:

* Patients with revision ACLR, bilateral ACLR, and postoperative infections were excluded from the study.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
KOOS | 1 week
  The primary variable of the study is the total KOOS score.

SECONDARY OUTCOMES:
Body mass index | 1 week
  Body mass (kg) and height (cm) were measured, and the body mass index (BMI) was calculated as kg/m2.
Oxford Knee Score (OKS) scoring | 1 week
  OKS consists of 12 questions. Standardized answer options are provided (5 Likert boxes), and each question is assigned a score from 0 to 4. A score of 40-48 indicates no symptoms or satisfactory joint function, 30-39 moderate knee arthritis, 20-29 moderate to severe knee arthritis, and 0-19 severe knee arthritis.
Tampa Scale of Kinesiophobia (TSK-17) | 1 week
  The Tampa Scale of Kinesiophobia (TSK-17) was developed as a self-reported checklist to measure fear of pain during movement and fear of reinjury. The TSK-17 consists of 17 questions. Standardized answer options are given as a 4-point Likert scale, and each question is assigned a score from 1 to 4. A normalized score between 17 and 68 points is calculated. A score of 37 or over indicates kinesiophobia.
Quadriceps and hamstring muscle isokinetic strength | 1 week
  Quadriceps and hamstring muscle strength at 60˚/s and 180˚/s were measured with an isokinetic dynamometer. For 180˚/s, five trial and fifteen testing repetitions were used, and for 60˚/s, three trial and three testing repetitions were used. The resting time between trial and testing was two minutes, between different speeds one minute, and between legs two minutes. The maximum peak torques were used in the statistical analysis.
Single-leg hop test | 1 week
  The single-leg hop test (SLHT) for distance was used for lower limb functional testing. The test started with the participant standing on one leg, toes behind a marked line, and hands on hips throughout to avoid aiding the jump by swinging the arms. The participant was instructed to jump as far as possible and land on the same leg without losing balance. If the patient made contact with the ground with the contralateral limb, lost balance, or made additional hops after landing, the distance was not measured and the jump void. The distance was measured from the starting line to the heel of the leg being tested. For both legs, three trials and three jumps for maximal effort were allowed. The longest distance for both the left leg and the right leg were used in the statistical analysis.
Y-balance test | 1 week
  The Y-balance test (YBT) (Move2Perform, United States) for anterior reach was used to measure dynamic balance. Participants performed three trials to familiarize themselves with the test, and then undertook three tests. The test started with the participant standing barefoot on the testing kit. The patients had to push a wooden box with the contralateral leg as far as possible with continuous movement and return to their starting position without losing balance. The longest distance achieved was used in the statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Leho Rips, MD, Principal Investigator — Tartu University Hospital
Locations (1):
- Tartu University Hospital, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rips L, Koovit T, Luik M, Saar H, Kuik R, Kartus JT, Rahu M. In the medium term, more than half of males report kinesiophobia after anterior cruciate ligament reconstruction. J ISAKOS. 2024 Oct;9(5):100309. doi: 10.1016/j.jisako.2024.100309. Epub 2024 Aug 17. PMID 39159822